CLINICAL TRIAL: NCT04095247
Title: Does Additional ECG-triggered Stimulation Increase the Efficacy of Vagus Nerve Stimulation? An Investigator-initiated Prospective, Multinational, Single Blinded, Randomized Cross-over Trial in Patients With VNS-treatment
Brief Title: Does Pulse-triggered VNS Autostimulation Increase VNS Efficacy
Acronym: ERAS
Status: Terminated | Type: Observational
Why Stopped: for few participants recruited
Sponsor: Oslo University Hospital (Other)
Collaborators: Filadelfia Epilepsy Hospital (Other); Rigshospitalet, Denmark (Other); Universitaire Ziekenhuizen KU Leuven (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Oliver Johannes Henning, Principal Investigator, Oslo University Hospital
Other Study IDs: 2018/667
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective

INTERVENTIONS:
Device: Vagus nerv stimulator — pulse triggered autostimulation

SUMMARY:
This is a research study to investigate whether the use of an extra function of vagus nerve stimulator (VNS) can give an improved effect against epilepsy. Many epileptic seizures are accompanied by an increase in heart rate. One auxiliary function of a new type of stimulator is continuous measurement of cardiac activity, and when pulse rate increases an extra stimulation is delivered. It has been shown that this can interrupt attacks that are about to develop. In this project the investigators will test how well that works for patients in daily life. The new type of stimulator has similar design and location as the old one. Patients who have already been treated with VNS and who need to switch the stimulator because the battery is starting to run out, are asked whether they want to participate. The study is a randomized and blinded cross-over. The activation of the extra feature is done either in the first or the second treatment phase. Which phase is the phase with activated autostimulation will be decided by random selection and the patient does not know when the auxiliary function is started. The study period is 11 months. Patients are asked to fill in some questionnaires on seizures, quality of life and quality of sleep.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, 12 years of age or older, who have a VNS without ECG-triggered auto stimulation implanted, have a positive effect and have a device replacement with model 106 or model 1000 due to low battery capacity,.
* Subjects, who have 2 or more seizure per month and not more than 28 days between seizures during the baseline.
* Subjects, who are on a stable regiment of antiepileptic drug treatment for at least 3 month prior to enrollment and maintain on this regimen throughout the study.
* VNS parameters have not been changed I the last 3 month prior to enrollment.
* Subjects which are using an off time of at least 1.8 min. (If the patient is on a duty cycle involving an off-time of 1.1 min. or less, and willing to participate in the study the duty cycle will have to be changed to fulfill the inclusion criteria as follows. The off-time will be changed to 1.8 min. and the on-time accordingly to achieve about the same duty cycle as the patient had before. If the duty cycle is above 30% the parameters will be changed to 60 sec./1.8 min., if the duty cycle is between 30% and 23% the parameters will be change to 30 sec./1,8 min., if the duty cycle is 20% the parameters will be change to 21 sec./1,8 min. and if the duty cycle is 15% the parameters will be change to 14 sec./1,8 min. After at periode of 3 month observation the patient can be included in the study.)
* Either the subjects or the legal guardian are able to agree to participate by signing the informed consent form.

Exclusion Criteria:

* Subjects with rapidly progressive neurodegenerative or rapidly progressing neoplastic disease.
* Subjects or legal guardians who are unable to understand the study procedures.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Eligible for the study are subjects (males and females) 12 years of age or older who had been using a VNS for at least three years with a positive effect and are getting a device replacement due to low battery capacity or who had a replacement and had not started the additional ECG -triggered stimulation before the study.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2022-04-06 (Actual); Study Completion 2022-04-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with >25 % change in seizure frequency | after 11 month
  Percentage of subjects with >25 % change in seizure frequency

SECONDARY OUTCOMES:
Change in mean National Hospital Seizure Severity Scale score | after 11 month
  Change in mean National Hospital Seizure Severity Scale score (range 1-22 Points, higher values indicate a worse situation)
Change in mean average seizure duration | after 11 month
  Change in mean average seizure duration

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Henning, MD, Principal Investigator — Oslo University Hospital
Locations (1):
- Norwegian epilepsy center, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No